CLINICAL TRIAL: NCT00418574
Title: A Randomised,Double Blind, Placebo Controlled, Multicentre Trial of Abagovomab Maintenance Therapy in Patients With Epithelial Ovarian Cancer After Complete Response to First Line Chemotherapy
Brief Title: Efficacy Multicentre Trial of ImmunoTherapy Vaccination With Abagovomab to Treat Ovarian Cancer Patients
Acronym: MIMOSA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No benefit on primary end point (RFS); no rationale to collect survival data
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABA-01; AGO-OVAR 10 (Other: AGO); 2006-002801-30 (EudraCT Number)
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Results first posted 2011-11-18 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Abagovomab
MeSH Terms: conditions — Ovarian Neoplasms | interventions — abagovomab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abagovomab (Experimental)
  Interventions: Biological: Abagovomab
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Abagovomab — 2 mg/ml SC (subcutaneously)
  Arms: Abagovomab
Biological: Placebo — 2 mg/ml SC (subcutaneously)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the benefit of vaccination with Abagovomab, an experimental immunotherapy in ovarian cancer patients. The benefit will be evaluated in terms of time the remission status is kept as well as prolongation of life expectancy.

DETAILED DESCRIPTION:
Standard initial treatment of ovarian cancer patients includes both surgery and chemotherapy which in the vast majority of cases achieves the disappearance of ovarian cancer lesions. This status, called "clinical remission" which means having no evidence of cancer on CT scan or physical examination needs to be carefully follow up in order to confirm the maintenance of the remission status or to early detect if the cancer grows again and then start a new chemotherapy. At present, no approved therapies exist for the maintenance treatment of patients who achieved the clinical remission.

This trial aims to evaluate if the repeated vaccination with Abagovomab creates an immunoresponse which is able to fight the cancer cells thus keeping the remission status as long as possible and help patients live disease-free and longer.

Patients who achieve the remission status after chemotherapy will be screened for study participation and if they meet the criteria for inclusion they will start to receive a single subcutaneous injection every 2 weeks (for the first 4 doses - induction phase) and then every 4 weeks (maintenance phase). The duration of treatment is up to approximately 4 years or it will be stopped in case relapse occurs.

In order to evaluate the real benefit of vaccination, the experimental treatment includes Abagovomab (the active drug) or placebo (the vehicle only, without drug), with a double chance to receive Abagovomab. Assignment of Abagovomab or placebo will be done by a computerised system and nobody in the study will know which treatment has been allocated until study end.

Patients will be visited every 4 weeks and will undergo CT scan of pelvis and abdomen every 12 weeks in order to confirm the remission status or to early detect if relapse eventually occurs. This will be done in blind condition (i.e. without being aware which treatment the patient is going to receive) for the first part of the study which is expected to last four years. After then the overall status of patient will continue to be monitored by phone contact for additional five years.

ELIGIBILITY:
Inclusion Criteria:

At a maximum of 12 weeks after the last cycle of first line standard platinum/taxane intravenous (IV) or intraperitoneal (IP) chemotherapy, patients must fulfill all the following inclusion criteria:

* Age >/= 18 years;
* Properly executed written informed consent;
* History of histological and CA125 (> 35 U/ml) confirmed diagnosis of stage III-IV epithelial ovarian, fallopian tube, or primary peritoneal cancer;
* History of debulking surgery and 6-8 cycles of standard platinum/taxane based non-investigational IV-IP chemotherapy;
* Complete clinical response defined as:
* Normal physical examination;
* No symptoms suggestive of persistent cancer;
* No definite evidence of disease by computed tomography (CT) of the abdomen and pelvis within the previous 4 weeks;
* Negative chest x-ray (or chest CT scan) within the previous 4 weeks;
* Serum CA125 within the normal laboratory range.
* Adequate hematologic, renal and hepatic function:

  * Absolute Neutrophil Count (ANC) >/=1.5 * 109/l;
  * Platelets >/= 75 * 109/l;
  * Haemoglobin >/= 6.2 mmol/l (>9.9 g/dl);
  * Serum creatinine </= 1.5 * ULN (Upper Limit of Normal);
  * Bilirubin </= 1.5 * ULN; AST, ALT, AP </= 2.5 * ULN.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) </= 2.

Exclusion Criteria:

Patients are ineligible to participate in the study, if any of the following criteria are present:

* any other invasive malignancies, with the exception of non-melanoma skin cancer or cervical carcinoma in situ, within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy;
* known active autoimmune disease requiring chronic treatment with immunosuppressive agents (e.g., rheumatoid arthritis, ulcerative colitis, etc.);
* known immune deficiency (e.g. HIV, hypogammaglobulinemia, etc.);
* known infection with hepatitis B, or hepatitis C;
* history of recent myocardial infarction (</= 6 months) or decompensated heart failure (New York Heart Association - NYHA class >/= III);
* previous or concomitant use of any anti-cancer therapy other than the platinum-taxane based 1st line chemotherapy for ovarian cancer; any maintenance or consolidation therapy is not permitted after completion of standard front line chemotherapy.
* concomitant use of any other investigational agent;
* any prior investigational anti-cancer vaccine or monoclonal antibody;
* known allergy to murine proteins;
* any significant medical or psychiatric condition, drug or alcohol abuse that might prevent the patient from complying with all study procedures;
* clinically significant active infection;
* concomitant use of any immunosuppressive agent (e.g., steroids, cyclosporin, etc.);
* major surgery within the previous 2 weeks;
* radiotherapy within the previous 4 weeks;
* any significant toxicity from prior chemotherapy;
* unreliability or inability to follow protocol requirements;
* potentially childbearing and not willing to use adequate contraceptive methods throughout the entire study period;
* pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 888 (Actual)
Dates: Start 2006-12; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacobus Pfisterer, MD, Study Chair — AGO-OVAR, Ovarian Cancer Study Group, Germany; Ubbo-Emmius-Klinik gGmbH Aurich, Germany; Paul Sabbatini, MD, Principal Investigator — Memorial Sloan-Kettering Cancer Centre- NY; Jonathan Berek, MD, Principal Investigator — COGI (Cooperative Ovarian Cancer Group for Immunotherapy); Dept Obstetrics and Gynecology, Stanford CA; Giovanni Scambia, MD, Principal Investigator — Universtita' Cattolica del Sacro Cuore, Dipartimento di Oncologia - Roma, Italy; Antonio Casado, MD, Principal Investigator — Hospital Clinico San Carlos, Servicio de Oncología Medica - Madrid, Spain; Anna Pluzanska, MD, Principal Investigator — Klinika Chemioterapii Nowotworów Akademii Medycznej w Łodzi, Regionalny Osrodek Onkologiczny - Lodz, Poland; Karel Cwiertka, MD, Principal Investigator — Onkologická klinika Fakultni Nemocnice Olomouc, Czech Republic; Tamás Pintér, MD, Principal Investigator — Petz Aladar Megyei Oktató Kórház, Onkoradiológia - Győr, Hungary; Eric Pujade-Lauraine, MD, Principal Investigator — Hôpital Hotel Dieu - Paris, France
Locations (150):
- United States (22):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Stanford University, Stanford, California
  - University of Colorado, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - University of Miami, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Curtis and Elizabeth Anderson Cancer Institute, Savannah, Georgia
  - Indiana University Cancer Pavilion, Indianapolis, Indiana
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - The Cancer Care Center, St Louis, Missouri
  - Women's Cancer Center, Las Vegas, Nevada
  - Hackensack University Medical Center, Obstetrics and Gynecology Oncology, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Centre, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - The West Clinic, Memphis, Tennessee
- Belgium (6):
  - Algemeen Stedelijk Ziekenhuis Aalst, Aalst
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent Medische Oncologie 4B-Z, Ghent
  - CHU de Liége (Sart Tilman), Liège
  - Clinique Sainte Elizabeth, Namur
  - AZ Sint Augustinus, Oncologisch Centrum GVA, Wilrijk
- Czechia (13):
  - Fakultni nemocnice Brno, Brno
  - MOU Zluty Kopec, Brno
  - Nemocnice Ceske Budejovice, a.s., České Budějovice
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Krajska nemocnice Liberec, oddeleni gynekologicko porodnicke, Liberec
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni Nemocnice Ostrava, Ostrava
  - Krajska nemocnice, Pardubice
  - Gynekologicko-porodnicka klinika FN Plzen, Pilsen
  - Fakultni nemocnice Královské Vinohrady, Prague
  - Vseobecna Fakultni Nemocnice, Prague
  - Fakultni nemocnice Bulovka, Prague
  - Krajska nemocnice T. Bati, Zlín
- France (4):
  - Institut Bergonié, Bordeaux
  - Centre Jean Bernard, Le Mans
  - Centre Catherine de Sienne, Nantes
  - Hôpital Hotel Dieu, Paris
- Germany (45):
  - Helios Kliniken GmbH, Klinikum Buch, Berlin
  - Charité - Campus Virchow Klinikum, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Bremen-Mitte gGmbH, Bremen
  - Klinikum Chemnitz GmbH, Chemnitz
  - St.-Josefs-Hospital Cloppenburg, Cloppenburg
  - Klinikum der Universität zu Köln, Cologne
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Evangelisches Krankenhaus, Düsseldorf
  - Kreisklinik Ebersberg gGmbH, Ebersberg
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum, Essen
  - Klinikum der JWG Universität Frankfurt, Frankfurt
  - Universitätsklinikum, Freiburg im Breisgau
  - Universitätsklinikum, Göttingen
  - Klinikum der Ernst-Moritz-Universität, Greifswald
  - Martin-Luther-Universität Halle-Wittenberg, Klinikum der Medizinischen Fakultät, Halle
  - Universitätskrankenhaus Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
  - St. Vincentius Kliniken AG, Karlsruhe
  - Klinikum Kassel, Kassel
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Kreiskrankenhaus Leonberg, Leonberg
  - Asklepios Klinik Lich, Lich
  - Vincenz-Krankenhaus, Limburg
  - Klinik St. Marienstift, Magdeburg
  - Städtisches Klinikum Magdeburg, Magdeburg
  - Otto-von-Guericke-Universität, Magdeburg
  - Johannes-Gutenberg-Universität, Mainz
  - Universitätsklinikum Gießen u. Marburg, Marburg
  - Klinikum der Universität München-Innenstadt, München
  - Klinikum Großhadern, München
  - Klinikum rechts der Isar, München
  - Klinikum Offenbach GmbH, Offenbach
  - St. Vincenz-Krankenhaus Paderborn, Paderborn
  - Elblandkliniken Meißen-Radebeul GmbH, Radebeul
  - Krankenhaus St. Josef, Regensburg
  - Klinikum Südstadt der Hansestadt Rostock, Rostock
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum, Ulm
  - Klinikum der Stadt Villingen-Schwenningen GmbH, Villingen-Schwenningen
  - St. Josefs-Hospital, Wiesbaden
  - r. Horst Schmidt Kliniken GmbH, Wiesbaden
  - Klinikum der Stadt Wolfsburg-FrauenklinikWolfsburg, Wolfsburg
- Hungary (8):
  - Fővárosi Önkormányzat Szent Margit Kórháza, Onkológia, Budapest
  - Semmelweis Egyetem II. sz. Szülészeti és Nőgyógyászati Klinika, Budapest
  - Semmelweis Egyetem, I sz. Szülészeti és Nőgyógyászati Klinika, Budapest
  - Debreceni Egyetem Orvos és Egészségtudományi Centrum, Szülészetl es Nőgyógyászatl Klinika, Debrecen
  - Petz Aladar Megyei Oktató Kórház, Onkoradiológia, Győr
  - Szabolcs-Szatmár-Bereg Megyei Önkormányzat Jósa András Kórháza, Szülészet-Nőgyógyászati Osztály, Nyíregyháza
  - Pécsi Tudományegyetem, ÁOK Szülészeti és Nőgyógyászati Klinika, Pécs
  - Komárom-Esztergom Megyei Onkormanyzat Szent Borbála Kórház, Szülészet-Nőgyógyászati Osztály, Tatabánya
- Italy (18):
  - Unità Operativa Ginecologia e Ostetricia 2^, Università degli studi di Bari, Policlinico, Bari
  - Ospedale S. Orsola Malpighi, Oncologia Medica, Bologna
  - Universtita' Cattolica del Sacro Cuore Dipartimento di Oncologia, Campobasso
  - DH Oncologico U.O. Medicina Oncologica Ospedale Ramazzini, Carpi (MO)
  - Oncologia Medica Ospedale di Faenza - AUSL di Ravenna, Faenza
  - Azienda Ospedaliera - Universitaria Careggi, Florence
  - Azienda Ospedaliera San Martino - Padiglione Malattie Complesse, Dipartimento di Oncologia Medica, Genova
  - Istituto Nazionale dei Tumori di Milano, Milan
  - Istituto Europeo di Oncologia - Divisione di Ginecologia, Milan
  - Policlinico di Modena, Dipartimento di Oncologia ed Ematologia, Modena
  - Istituto Nazionale per lo studio e la cura dei tumori "Fondazione Pascale" Oncologia Medica, Napoli
  - Azienda Ospedaliera San Carlo - Oncologia Medica, Potenza
  - Ospedali Riuniti Bianchi-Melacrino-Morelli - Oncologia Medica, Reggio Calabria
  - Arcispedale Santa Maria Nuova, Oncologia Medica, Reggio Emilia
  - Policlinico Umberto I D.H. Oncologico Oncologia Medica, Roma
  - Dipartimento di Ginecologia ed Ostetricia Policlinico Universitario Gemelli, Roma
  - Ospedale Casa Sollievo della Sofferenza - Unita' Operativa di Ostetricia e Ginecologia, San Giovanni Rotondo (FG)
  - Dipartimento di Discipline Ginecologiche e Ostetriche - Universita degli Studi di Torino - Azienda ospedaliera O.I.R.M.-S'Anna, Torino
- Poland (13):
  - Wojewódzki Szpital Specjalistyczny Nr 4, Bytom
  - Oddzial Onkologii Wojewódzki Szpital Specjalistyczny, Częstochowa
  - Wojewodzkie Centrum Onkologii, Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Gdansk
  - Vesalius Kraków, Krakow
  - "Centrum Onkologii, Instytut im. M. Skłodowskiej-Curie, Oddział w Krakowie,, Krakow
  - Klinika Chemioterapii Nowotworów Akademii Medycznej w Łodzi, Regionalny Osrodek Onkologiczny, Lodz
  - Oddzial Chemioterapii ZOZ MSWiA z Warminsko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - Klinika Onkologii, Oddzial Chemioterapii Akademii Medycznej w Poznaniu, Poznan
  - SPZOZ Wojewodzki Szpital Specjalistyczny Nr 3, Oddzial Onkologii, Rybnik
  - Wojewodzki Szpital Zespolony, Oddzial Onkologii Klinicznej, Torun
  - Wojskowy Instytut Medyczny; Klinika Onkologii Centralnego Szpitala Klinicznego MON, Warsaw
  - Centralny Szpital Kliniczny MSWiA, Klinika Onkologii, Hematologii i Chorob Wewnetrznych, Warsaw
  - Centrum Onkologii Instytut im. Marii Sklodowskiej-Curie, Klinika Nowotworów Narządów Płciowych Kobiecych, Warsaw
- Spain (21):
  - Centro Oncológico Regional de Galicia, Servicio de Oncologia Medica, A Coruña
  - Hospital Germans Trias y Pujol, Badalona
  - Hospital Vall d'Hebrón, Servicio de Oncologia, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Servicio de Oncologia, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital de Elche, Servico de Oncologia, Elche
  - Instituto Catalán de Oncología - Hospital Universitari de Girona "Dr. Josep Trueta". Oncologia Medica, Girona
  - Hospital Virgen de las Nieves, Granada
  - Hospital Juan Ramón Jiménez de Huelva, Huelva
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario Arnau de Vilanova, Servicio de Oncologia, Lleida
  - MD Anderson Internacional Espana, Madrid
  - Hospital Clinico San Carlos, Servicio de Oncología Medica, Madrid
  - Hospital de Mataró, Mataró
  - Hospital Clinico de Malaga. Servicio de Oncologia, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Son Dureta, Servicio de Oncología, Palma de Mallorca
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital General Universitario de Valencia, Valencia

REFERENCES:
- [Background] Reinartz S, Kohler S, Schlebusch H, Krista K, Giffels P, Renke K, Huober J, Mobus V, Kreienberg R, DuBois A, Sabbatini P, Wagner U. Vaccination of patients with advanced ovarian carcinoma with the anti-idiotype ACA125: immunological response and survival (phase Ib/II). Clin Cancer Res. 2004 Mar 1;10(5):1580-7. doi: 10.1158/1078-0432.ccr-03-0056. PMID 15014007
- [Background] Wagner U, Kohler S, Reinartz S, Giffels P, Huober J, Renke K, Schlebusch H, Biersack HJ, Mobus V, Kreienberg R, Bauknecht T, Krebs D, Wallwiener D. Immunological consolidation of ovarian carcinoma recurrences with monoclonal anti-idiotype antibody ACA125: immune responses and survival in palliative treatment. See The biology behind: K. A. Foon and M. Bhattacharya-Chatterjee, Are solid tumor anti-idiotype vaccines ready for prime time? Clin. Cancer Res., 7:1112-1115, 2001. Clin Cancer Res. 2001 May;7(5):1154-62. PMID 11350879
- [Background] Pfisterer J, du Bois A, Sehouli J, Loibl S, Reinartz S, Reuss A, Canzler U, Belau A, Jackisch C, Kimmig R, Wollschlaeger K, Heilmann V, Hilpert F. The anti-idiotypic antibody abagovomab in patients with recurrent ovarian cancer. A phase I trial of the AGO-OVAR. Ann Oncol. 2006 Oct;17(10):1568-77. doi: 10.1093/annonc/mdl357. PMID 17005631
- [Background] Sabbatini P, Dupont J, Aghajanian C, Derosa F, Poynor E, Anderson S, Hensley M, Livingston P, Iasonos A, Spriggs D, McGuire W, Reinartz S, Schneider S, Grande C, Lele S, Rodabaugh K, Kepner J, Ferrone S, Odunsi K. Phase I study of abagovomab in patients with epithelial ovarian, fallopian tube, or primary peritoneal cancer. Clin Cancer Res. 2006 Sep 15;12(18):5503-10. doi: 10.1158/1078-0432.CCR-05-2670. PMID 17000686
- [Derived] Buzzonetti A, Fossati M, Catzola V, Scambia G, Fattorossi A, Battaglia A. Immunological response induced by abagovomab as a maintenance therapy in patients with epithelial ovarian cancer: relationship with survival-a substudy of the MIMOSA trial. Cancer Immunol Immunother. 2014 Oct;63(10):1037-45. doi: 10.1007/s00262-014-1569-0. Epub 2014 Jun 21. PMID 24952307
- [Derived] Sabbatini P, Harter P, Scambia G, Sehouli J, Meier W, Wimberger P, Baumann KH, Kurzeder C, Schmalfeldt B, Cibula D, Bidzinski M, Casado A, Martoni A, Colombo N, Holloway RW, Selvaggi L, Li A, del Campo J, Cwiertka K, Pinter T, Vermorken JB, Pujade-Lauraine E, Scartoni S, Bertolotti M, Simonelli C, Capriati A, Maggi CA, Berek JS, Pfisterer J. Abagovomab as maintenance therapy in patients with epithelial ovarian cancer: a phase III trial of the AGO OVAR, COGI, GINECO, and GEICO--the MIMOSA study. J Clin Oncol. 2013 Apr 20;31(12):1554-61. doi: 10.1200/JCO.2012.46.4057. Epub 2013 Mar 11. PMID 23478059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study population was recruited in 139 sites (Hospitals/University Clinics) distributed in Europe (Belgium, Czech Republic, France, Germany, Hungary, Italy, Poland and Spain) and US.
  Date of first patient randomised: 08 December 2006 Date of last patient randomised: 26 December 2008
Groups:
- Abagovomab; Placebo: 2 mg/ml SC, every 2 weeks (for the first 4 doses - induction phase) and then every 4 weeks (maintenance phase)
Period: Overall Study
Arm/Group | Abagovomab | Placebo
Started | 593 | 295
TREATED | 592 | 294
Completed | 545 | 272
Not Completed | 48 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abagovomab | Placebo | Total
Number analyzed (Participants) | 593 | 295 | 888
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 447 | 227 | 674
  >=65 years | 145 | 68 | 213
Age Continuous [Mean (Standard Deviation); unit: years] | 56.4 (10.57) | 56.0 (10.47) | 56.3 (10.53)
Sex/Gender, Customized [Number; unit: participants]
  Female | 593 | 295 | 888
Region of Enrollment [Number; unit: participants]
  France | 1 | 2 | 3
  United States | 91 | 47 | 138
  Hungary | 17 | 8 | 25
  Czech Republic | 54 | 28 | 82
  Poland | 53 | 25 | 78
  Spain | 55 | 48 | 103
  Belgium | 19 | 4 | 23
  Germany | 206 | 93 | 299
  Italy | 97 | 40 | 137
Histology of ovarian tumor [Number; unit: participants]
  Serous/papillary | 481 | 245 | 726
  Endometrioid | 38 | 21 | 59
  Mucinous | 6 | 3 | 9
  Undifferentiated | 14 | 7 | 21
  Mixed tumor | 18 | 7 | 25
  Others | 33 | 12 | 45
  missing | 3 | 0 | 3
Eastern Cooperative Oncology Group Performance Status (ECOG-PS) [Number; unit: participants] — This scale and criteria are used by doctors and researchers to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis. The scale runs from the score 0 to 5, with 0 denoting the status "Fully active, able to carry on all pre-disease performance without restriction" and 5 the status "Dead".
  participants
    0 | 460 | 240 | 700
    1 | 131 | 55 | 186
    2 | 2 | 0 | 2
Grade of histologic differentiation [Number; unit: participants] — Histologic grade, also called differentiation, refers to how much the tumor cells resemble normal cells of the same tissue type.
  GX Grade cannot be assessed (Undetermined grade) G1 Well-differentiated (Low grade) - best prognosis G2 Moderately differentiated (Intermediate grade) G3 Poorly differentiated (High grade) G4 Undifferentiated (High grade) - worst prognosis
  participants
    G1-G2 | 160 | 82 | 242
    G3-G4 | 365 | 185 | 550
    GX | 12 | 4 | 16
    not done | 56 | 24 | 80
International Federation of Gynecology and Obstetrics (FIGO) stage [Number; unit: participants] — International system of staging which identifies the spread of the ovarian cancer at the point of diagnosis [STAGE 1 - Tumour is confined to the ovary / ovaries; STAGE 2 - Tumour involves one or both ovaries and has extended into the pelvis; STAGE 3 - The tumour involves one or both ovaries with microscopically confirmed peritoneal metastasis outside the pelvis and/or regional lymph node metastasis, includes liver capsule metastasis; STAGE: 4 - Distant metastasis beyond the peritoneal cavity, liver parenchymal metastasis.]
  participants
    III | 513 | 252 | 765
    IV | 80 | 42 | 122
    missing | 0 | 1 | 1
Tumor size after debulking surgery [Number; unit: participants]
  <= 1 cm | 479 | 232 | 711
  > 1 cm | 114 | 63 | 177
Serum CA-125 after 3rd chemotherapy cycle [Number; unit: participants]
  <= 35 U/ml | 479 | 239 | 718
  > 35 U/ml | 114 | 55 | 169
  missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Free Survival Evaluated by Clinical Event Adjudication Committee (CEAC)
Description: The Recurrence free survival correspond to the time from date of randomization to documented disease recurrence or death. Disease recurrence is defined as the appearance of any lesion or development of tumor-related symptoms evaluated by medical examination and must be confirmed by a documented CT scan.
Time Frame: Every 12 weeks up to recurrence or up to 3 months after last administered dose
Population: intention to treat (ITT) population (i.e. all randomized patients)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Abagovomab | Placebo
Number analyzed (Participants) | 593 | 295
days | 403 [323 to 414] | 402 [323 to 487]
Statistical Analysis 1: Comparison: Abagovomab vs Placebo; Test type: Superiority or Other; p = 0.301, Regression, Cox; Hazard Ratio (HR) = 1.099, 95% CI 2-sided [0.919 to 1.315]

2. Secondary Outcome: Overall Survival
Description: 2 years survival rate
Time Frame: 2 years
Population: intention to treat (ITT) population (i.e. all randomized patients)
Measure: Number; unit: Percentage of participants
Arm/Group | Abagovomab | Placebo
Number analyzed (Participants) | 593 | 295
Percentage of participants | 80 | 79

3. Secondary Outcome: Safety
Description: Safety was analyzed in all patients who received at least 1 dose administration.
  Adverse event (AE) are defined as events which started on or after the first dose of study medication and on or before the date of the final study visit, or within 12 weeks of the last dose if the final study visit was not performed.
Time Frame: Along treatment administration and up to double blind observation period. i.e. for each patient after the first dose administration till the f inal study visit, or within 12 weeks of the last dose
Population: Safety population (i.e. All randomized patients who received at least one dose treatment administration)
Measure: Number; unit: participants
Arm/Group | Abagovomab | Placebo
Number analyzed (Participants) | 592 | 294
participants
  Patients with at least 1 Adverse Event (AE) | 564 | 278
  Patients with at least 1 Adverse Drug Reaction ADR | 507 | 246
  Patients with at least 1 Serious Adverse Event SAE | 141 | 72
  Patients with at least 1 Serious ADR (SADR) | 10 | 3
  Patients with at least 1 AE leading to withdrawal | 93 | 57
  Patients with at least 1 AE resulted in death | 8 | 4

4. Secondary Outcome: Time Course of Immunoresponse
Description: Time course of immunologic parameters (anti-anti-idiotypic antibody - Ab3) will be assessed in all patients, by comparing levels at baseline (week 0), at week 10 after first dose administration and at end of treatment (at week 4 or week 12 after the last administered dose, as appropriate).
Time Frame: at baseline, at week 10 after first dose administration and at final study visit (at week 4 or week 12 after the last administered dose, as appropriate)
Population: Participants who received abagovomab (evaluable population)and have baseline serum sample: 576 at baseline; 538 at week 10 after first dose intake; 449 at the final study visit
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Abagovomab
Number analyzed (Participants) | 576
ng/ml
  Ab3 (baseline) | 0 [0 to 118000]
  Ab3 (week 10) | 63550 [0 to 777000]
  Ab3 (end of treatment) | 493000 [0 to 2720000]

ADVERSE EVENTS:
Time Frame: 4 years
Description: Adverse Events monitored throughout the observation period, at each visit prior dosing (every 2 weeks during the induction phase, every 4 weeks during the maintenance phase)
Arm/Group | Abagovomab | Placebo
Serious Adverse Events (participants affected / at risk) | 141/592 | 72/294
Other Adverse Events (participants affected / at risk) | 532/592 | 261/294
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abagovomab (N=592) | Placebo (N=294)
Anaemias NEC (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphatic system disorders NEC (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenias (Blood and lymphatic system disorders) | 1 (6) | 0 (0)
Ischaemic coronary artery disorders (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial disorders NEC (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular arrhythmias (Cardiac disorders) | 1 (2) | 0 (0)
Inner ear signs and symptoms (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane disorders (excl infections) (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Thyroid disorders NEC (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid hyperfunction disorders (Endocrine disorders) | 0 (0) | 1 (2)
Glaucomas (excl congenital) (Eye disorders) | 1 (1) | 0 (0)
Retinal structural change, deposit and degeneration (Eye disorders) | 0 (0) | 1 (1)
Abdominal findings abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernias, site unspecified (Gastrointestinal disorders) | 1 (1) | 4 (4)
Acute and chronic pancreatitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Diarrhoea (excl infective) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal and small intestinal stenosis and obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dyspeptic signs and symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric and oesophageal haemorrhages (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (excl infective) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal and abdominal pains (excl oral and throat) (Gastrointestinal disorders) | 11 (13) | 4 (4)
Gastrointestinal atonic and hypomotility disorders NEC (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrointestinal inflammatory disorders NEC (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal necrosis and gangrene (excl gangrenous hernia) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal stenosis and obstruction NEC (Gastrointestinal disorders) | 14 (15) | 12 (17)
Large intestinal stenosis and obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea and vomiting symptoms (Gastrointestinal disorders) | 3 (5) | 4 (5)
Non-site specific gastrointestinal haemorrhages (Gastrointestinal disorders) | 2 (2) | 1 (1)
Peritoneal and retroperitoneal disorders (Gastrointestinal disorders) | 18 (22) | 6 (6)
Peritoneal and retroperitoneal fibrosis and adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Device issues NEC (General disorders) | 0 (0) | 1 (1)
Febrile disorders (General disorders) | 3 (3) | 2 (3)
General signs and symptoms NEC (General disorders) | 3 (3) | 0 (0)
Hernias NEC (General disorders) | 2 (2) | 2 (2)
Injection site reactions (General disorders) | 0 (0) | 1 (1)
Oedema NEC (General disorders) | 2 (2) | 0 (0)
Pain and discomfort NEC (General disorders) | 2 (2) | 1 (1)
Therapeutic and nontherapeutic responses (General disorders) | 1 (1) | 0 (0)
Cholecystitis and cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholestasis and jaundice (Hepatobiliary disorders) | 1 (1) | 1 (2)
Gallbladder disorders NEC (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic conditions NEC (Immune system disorders) | 1 (1) | 0 (0)
Abdominal and gastrointestinal infections (Infections and infestations) | 2 (2) | 2 (2)
Aspergillus infections (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infections NEC (Infections and infestations) | 0 (0) | 1 (1)
Dental and oral soft tissue infections (Infections and infestations) | 0 (0) | 1 (1)
Ear infections (Infections and infestations) | 1 (1) | 0 (0)
Herpes viral infections (Infections and infestations) | 0 (0) | 2 (2)
Influenza viral infections (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract and lung infections (Infections and infestations) | 0 (0) | 1 (1)
Sepsis, bacteraemia, viraemia and fungaemia NEC (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal infections (Infections and infestations) | 1 (1) | 3 (4)
Upper respiratory tract infections (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infections (Infections and infestations) | 3 (3) | 0 (0)
Vascular infections (Infections and infestations) | 1 (1) | 0 (0)
Abdominal injuries NEC (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lower limb fractures and dislocations (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Non-site specific injuries NEC (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Non-site specific procedural complications (Injury, poisoning and procedural complications) | 7 (8) | 0 (0)
Pelvic fractures and dislocations (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Spinal fractures and dislocations (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Upper limb fractures and dislocations (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Digestive enzymes (Investigations) | 1 (2) | 0 (0)
Liver function analyses (Investigations) | 3 (5) | 0 (0)
Renal function analyses (Investigations) | 2 (2) | 0 (0)
Skeletal and cardiac muscle analyses (Investigations) | 1 (2) | 0 (0)
Tissue enzyme analyses NEC (Investigations) | 1 (1) | 0 (0)
Appetite disorders (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (incl subtypes) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bone related signs and symptoms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc disorders NEC (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint related signs and symptoms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Metabolic bone disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue pain and discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthropathies (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Soft tissue disorders NEC (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spine and neck deformities (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone neoplasms benign (excl cysts) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endocrine neoplasms malignant and unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal neoplasms malignant NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to specified sites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (16) | 13 (13)
Neoplasms malignant site unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasms unspecified malignancy and site unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Nervous system neoplasms unspecified malignancy NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell neoplasms malignant of the respiratory tract cell type specified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oncologic complications and emergencies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ovarian neoplasms malignant (excl germ cell) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 61 (80) | 41 (46)
Rectal neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin neoplasms malignant and unspecified (excl melanoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vaginal neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central nervous system haemorrhages and cerebrovascular accidents (Nervous system disorders) | 3 (3) | 1 (1)
Disturbances in consciousness NEC (Nervous system disorders) | 0 (0) | 1 (1)
Neurological signs and symptoms NEC (Nervous system disorders) | 2 (2) | 1 (1)
Peripheral neuropathies NEC (Nervous system disorders) | 0 (0) | 1 (1)
Seizures and seizure disorders NEC (Nervous system disorders) | 2 (2) | 0 (0)
Speech and language abnormalities (Nervous system disorders) | 0 (0) | 1 (1)
Transient cerebrovascular events (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety symptoms (Psychiatric disorders) | 1 (1) | 0 (0)
Depressive disorders (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure and impairment (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal obstructive disorders (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureteric disorders NEC (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast disorders NEC (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic prolapse conditions (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine disorders NEC (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breathing abnormalities (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumothorax and pleural effusions NEC (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 5 (5)
Pulmonary thrombotic and embolic conditions (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Connective tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal and epidermal conditions NEC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis and eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Accelerated and malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
Aortic embolism and thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Lymphangiopathies (Vascular disorders) | 3 (6) | 0 (0)
Lymphoedemas (Vascular disorders) | 0 (0) | 1 (1)
Non-site specific embolism and thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Peripheral embolism and thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abagovomab (N=592) | Placebo (N=294)
Diarrhoea (excl infective) (Gastrointestinal disorders) | 98 (177) | 41 (64)
Flatulence, bloating and distension (Gastrointestinal disorders) | 45 (69) | 25 (33)
Gastrointestinal and abdominal pains (excl oral and throat) (Gastrointestinal disorders) | 183 (300) | 81 (125)
Gastrointestinal atonic and hypomotility disorders NEC (Gastrointestinal disorders) | 82 (115) | 38 (54)
Nausea and vomiting symptoms (Gastrointestinal disorders) | 130 (325) | 64 (138)
Asthenic conditions (General disorders) | 191 (431) | 89 (240)
Febrile disorders (General disorders) | 67 (111) | 40 (73)
Feelings and sensations NEC (General disorders) | 34 (42) | 14 (25)
General signs and symptoms NEC (General disorders) | 44 (75) | 19 (25)
Injection site reactions (General disorders) | 467 (4906) | 222 (2352)
Oedema NEC (General disorders) | 61 (82) | 32 (39)
Pain and discomfort NEC (General disorders) | 37 (44) | 20 (22)
Lower respiratory tract and lung infections (Infections and infestations) | 43 (49) | 8 (8)
Upper respiratory tract infections (Infections and infestations) | 142 (242) | 70 (124)
Urinary tract infections (Infections and infestations) | 80 (114) | 27 (33)
Physical examination procedures (Investigations) | 33 (46) | 20 (33)
Bone related signs and symptoms (Musculoskeletal and connective tissue disorders) | 41 (59) | 26 (44)
Joint related signs and symptoms (Musculoskeletal and connective tissue disorders) | 134 (263) | 67 (112)
Muscle pains (Musculoskeletal and connective tissue disorders) | 59 (104) | 35 (59)
Musculoskeletal and connective tissue pain and discomfort (Musculoskeletal and connective tissue disorders) | 171 (355) | 79 (212)
Headaches NEC (Nervous system disorders) | 83 (227) | 38 (86)
Neurological signs and symptoms NEC (Nervous system disorders) | 42 (63) | 25 (30)
Peripheral neuropathies NEC (Nervous system disorders) | 46 (57) | 25 (28)
Disturbances in initiating and maintaining sleep (Psychiatric disorders) | 31 (37) | 17 (24)
Bladder and urethral symptoms (Renal and urinary disorders) | 38 (47) | 25 (30)
Breathing abnormalities (Respiratory, thoracic and mediastinal disorders) | 48 (59) | 23 (26)
Coughing and associated symptoms (Respiratory, thoracic and mediastinal disorders) | 43 (51) | 25 (31)
Erythemas (Skin and subcutaneous tissue disorders) | 40 (76) | 22 (37)
Pruritus NEC (Skin and subcutaneous tissue disorders) | 30 (50) | 15 (16)
Rashes, eruptions and exanthems NEC (Skin and subcutaneous tissue disorders) | 33 (47) | 19 (23)
Peripheral vascular disorders NEC (Vascular disorders) | 49 (62) | 26 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that result communications shall be exchanged and discussed with the sponsor 60 days prior to submission for publication or presentation.